CLINICAL TRIAL: NCT01642251
Title: Phase I and Randomized Phase II Double Blind Clinical Trial of Cisplatin and Etoposide in Combination With Veliparib (ABT-888) or Placebo as Frontline Therapy for Extensive Stage Small Cell Lung Cancer
Brief Title: Cisplatin and Etoposide With or Without Veliparib in Treating Patients With Extensive Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-01985; E2511 (Other: ECOG-ACRIN Cancer Research Group); U10CA180820 (NIH); U10CA021115 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Extensive Stage Small Cell Lung Carcinoma; Large Cell Lung Carcinoma; Neuroendocrine Carcinoma; Small Cell Carcinoma; Stage IV Non-Small Cell Lung Cancer AJCC v7
Keywords: Veliparib; Small cell lung cancer
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Carcinoma, Small Cell; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Cisplatin; Platinum; Etoposide; Podophyllotoxin; veliparib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (veliparib) (Experimental): Patients receive veliparib PO BID on days 1-7, etoposide IV over 60-120 minutes on days 1-3, and cisplatin IV over 60-120 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Etoposide; Drug: Veliparib
- Arm B (placebo) (Active Comparator): Patients receive placebo PO BID on days 1-7, etoposide IV over 60-120 minutes on days 1-3, and cisplatin IV over 60-120 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Etoposide; Drug: Placebo

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Cisdiaminedichloroplatinum; Cis -diaminedichloroplatinum (II); diaminedichloroplatinum; Platinol -AQ; Cis-platinum; P latinol; platinum; DDP; CDDP; DACP; NSC 119875
Drug: Etoposide — Given IV
  Other Names: Epipodophyllotoxin; EPEG; Vepesid; VP 16-213; VP-16
Drug: Veliparib — Given PO
  Other Names: ABT-888; PARP-1 inhibitor ABT-888; A-861695.0
  Arms: Arm A (veliparib)
Drug: Placebo — placebo of Veliparib
  Other Names: placebo therapy
  Arms: Arm B (placebo)

SUMMARY:
This randomized phase I/II trial studies the side effects and best dose of veliparib when given together with or without cisplatin and etoposide and to see how well they work in treating patients with extensive stage small cell lung cancer or large cell neuroendocrine non-small cell lung cancer that has spread to other parts of the body. Drugs used in chemotherapy, such as cisplatin and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving cisplatin and etoposide with or without veliparib may work better in treating patients with extensive stage small cell lung cancer or metastatic large cell neuroendocrine non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose (RP2D) of veliparib to use in combination with cisplatin and etoposide (CE). (Phase I) II. To determine whether the addition of ABT-888 (veliparib) to cisplatin etoposide (CE) results in improved progression free survival (PFS) over CE with placebo in the frontline therapy of newly diagnosed extensive stage small cell lung cancer. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the overall survival (OS) associated with the combination of CE plus ABT-888. (Phase II) II. To assess the overall response rate (ORR) as well as complete response rate (CRR) associated with the combination of CE plus ABT-888. (Phase II) III. To determine the toxicity profile of the combination of ABT-888 and CE chemotherapy in this patient population. (Phase II)

OTHER PRE-SPECIFIED OBJECTIVES:

I. To conduct exploratory correlative analysis of the impact of the select biomarkers. (Phase II) II. To compare the overall toxicity profile and specifically the incidence and severity of chemotherapy-induced peripheral neuropathy with the addition of ABT-888 to CE. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of veliparib followed by a phase II study.

Phase I: Patients receive veliparib orally (PO) twice daily (BID) on days 1-7, etoposide intravenously (IV) over 60-120 minutes on days 1-3, and cisplatin IV over 60-120 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Phase II: Patients are randomized to 1 of 2 treatment arms.

ARM D: Patients receive veliparib PO BID on days 1-7, etoposide IV over 60-120 minutes on days 1-3, and cisplatin IV over 60-120 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

ARM E: Patients receive placebo PO BID on days 1-7, etoposide IV over 60-120 minutes on days 1-3, and cisplatin IV over 60-120 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 1 year.

ELIGIBILITY:
PHASE I

Inclusion Criteria (phase I):

* Women must not be pregnant or breastfeeding; breastfeeding must be discontinued or the subject is not eligible for the study
* All females of childbearing potential must have a blood test within 2 weeks prior to randomization to rule out pregnancy; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception
* Patients must have histologically or cytologically confirmed:

  * Extensive stage small cell lung cancer (SCLC) or
  * Stage IV (M1a or M1b according to American Joint Committee on Cancer [AJCC] Staging Manual, 7th edition) large cell neuroendocrine non-small cell lung cancer (NSCLC) or
  * Small cell carcinoma of unknown primary or extrapulmonary origin and must be a candidate for systemic therapy

    * NOTE: The extensive disease SCLC classification for this protocol includes all patients with disease sites not defined as limited stage; limited stage disease category includes patients with disease restricted to one hemithorax with regional lymph node metastases, including hilar, ipsilateral and contralateral mediastinal, and/or ipsilateral supraclavicular nodes; extensive disease patients are defined as those patients with extrathoracic metastatic disease, malignant pleural effusion, bilateral or contralateral supraclavicular adenopathy
* Patients must have measurable or non-measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; baseline measurements and evaluations of all sites of disease must be obtained =< 4 weeks prior to registration (Phase I)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Absolute neutrophil count >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Leukocytes >= 3,000/mm^3
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 times institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase[SGPT]) =< 3 times institutional ULN (=< 5 times if liver function test [LFT] elevations due to known liver metastases)
* Creatinine =< 1.5 X ULN OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels > 1.5 x ULN
* Patients with central nervous system (CNS) metastases or a history of CNS metastases are ineligible
* Patients cannot have had prior chemotherapy or biologic therapy for SCLC or large cell neuroendocrine NSCLC, or small cell carcinoma of unknown primary or extrapulmonary origin; patients receiving prior radiation cannot register within 7 days after completion of radiation, and must have resolved adverse events attributed to radiation to =< grade 1; no previous irradiation to the only site of measurable or evaluable disease, unless that site had subsequent evidence of progression
* Patients receiving prior radiation cannot register within 7 days after completion of radiation, and must have resolved adverse events attributed to radiation to =< grade 1; no previous irradiation to the only site of measurable or evaluable disease, unless that site had subsequent evidence of progression
* Patients must NOT have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patient must be able to swallow pills

Exclusion Criteria (phase I):

* Patients have active seizure(s) or history of seizure(s)
* Patients have history of allergic reactions attributed to compounds of similar chemical or biologic composition to veliparib or other agents used in the study

PHASE II

Inclusion Criteria (phase II):

* Women must not be pregnant or breastfeeding; breastfeeding must be discontinued or the subject is not eligible for the study
* All females of childbearing potential must have a blood test within 2 weeks prior to randomization to rule out pregnancy; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months) with the current month counted as month 1
* Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception
* Patients must have extensive stage, histologically or cytologically confirmed small cell lung cancer; NOTE: the extensive disease classification for this protocol includes all patients with disease sites not defined as limited stage; limited stage disease category includes patients with disease restricted to one hemithorax with regional lymph node metastases, including hilar, ipsilateral and contralateral mediastinal, and/or ipsilateral supraclavicular nodes; extensive disease patients are defined as those patients with extrathoracic metastatic disease, malignant pleural effusion, bilateral or contralateral supraclavicular adenopathy
* Patients must have measurable disease based on RECIST 1.1; baseline measurements and evaluations of all sites of disease must be obtained =< 4 weeks prior to registration
* ECOG performance status 0 or 1
* Absolute neutrophil count >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Leukocytes >= 3,000/mm^3
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 times institutional upper limit of normal (ULN)
* AST (SGOT) and ALT (SGPT) =< 3 times institutional ULN (=< 5 times if LFT elevations due to known liver metastases)
* Creatinine =< 1.5 X ULN OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels > 1.5 x ULN
* Patients cannot have had prior chemotherapy or biologic therapy for small cell lung cancer; patients receiving prior radiation cannot register within 7 days after completion of radiation, and must have resolved adverse events attributed to radiation to =< grade 1; no previous irradiation to the only site of measurable or evaluable disease, unless that site had subsequent evidence of progression
* Patient must be able to swallow pills
* Patients may not be receiving any other investigational agents while on study

Exclusion Criteria (phase II):

* Patients with CNS metastases or a history of CNS metastases are ineligible
* Patients have history of allergic reactions attributed to compounds of similar chemical or biologic composition to veliparib or other agents used in the study
* Patients have active seizure(s) or history of seizure(s)
* Patients must NOT have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with veliparib; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2012-09-28; Primary Completion 2016-12-08 (Actual); Study Completion 2018-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taofeek Owonikoko, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (428):
- United States (428):
  - Loma Linda University Medical Center, Loma Linda, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - NorthShore Hematology Oncology-Libertyville, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Michiana Hematology Oncology PC-Crown Point, Crown Point, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Urology Cancer Center PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center-Manchester, Manchester, New Hampshire
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Geisinger Medical Oncology-Pottsville, Pottsville, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Kingsport, Kingsport, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Saint Clare's Hospital, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Result] Owonikoko TK, Dahlberg SE, Sica GL, Wagner LI, Wade JL 3rd, Srkalovic G, Lash BW, Leach JW, Leal TB, Aggarwal C, Ramalingam SS. Randomized Phase II Trial of Cisplatin and Etoposide in Combination With Veliparib or Placebo for Extensive-Stage Small-Cell Lung Cancer: ECOG-ACRIN 2511 Study. J Clin Oncol. 2019 Jan 20;37(3):222-229. doi: 10.1200/JCO.18.00264. Epub 2018 Dec 5. PMID 30523756
- [Derived] Steffen McLouth LE, Zhao F, Owonikoko TK, Feliciano JL, Mohindra NA, Dahlberg SE, Wade JL 3rd, Srkalovic G, Lash BW, Leach JW, Leal TA, Aggarwal C, Cella D, Ramalingam SS, Wagner LI. Patient-reported tolerability of veliparib combined with cisplatin and etoposide for treatment of extensive stage small cell lung cancer: Neurotoxicity and adherence data from the ECOG ACRIN cancer research group E2511 phase II randomized trial. Cancer Med. 2020 Oct;9(20):7511-7523. doi: 10.1002/cam4.3416. Epub 2020 Aug 28. PMID 32860331
- See also: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive." — https://nctn-data-archive.nci.nih.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened to accrual on 9/28/2012, was suspended to accrual on 7/23/2013 after nine patients had been enrolled to phase I portion of the trial (3 patients at dose level 1; 6 patients at dose level 2). Phase II portion of the trial was activated on 10/24/2013 and enrolled 147 patients prior to study accrual completion on 7/2/2015.
Groups:
- Phase I: Arm A (Dose Level 1); Phase I: Arm B (Dose Level II): The phase I portion of the study was designed to determine the recommended dose for veliparib for the phase II portion of the trial. A total of 9 patients were treated on the phase I study. A total of 3 dose levels of veliparib were planned: 60mg (level 1), 100gm (level 2) and 40mg (level -1). 1 cycle=3 weeks, maximum of 4 cycles.
- Phase II: Arm D (Veliparib): Patients receive veliparib PO BID on days 1-7, etoposide IV over 60-120 minutes on days 1-3, and cisplatin IV over 60-120 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Cisplatin: Given IV
  Etoposide: Given IV
  Veliparib: Given PO
- Phase II: Arm E (Placebo): Patients receive placebo PO BID on days 1-7, etoposide IV over 60-120 minutes on days 1-3, and cisplatin IV over 60-120 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Cisplatin: Given IV
  Etoposide: Given IV
  Placebo: placebo of Veliparib
Period: Overall Study
Arm/Group | Phase I: Arm A (Dose Level 1) | Phase I: Arm B (Dose Level II) | Phase II: Arm D (Veliparib) | Phase II: Arm E (Placebo)
Started | 3 | 6 | 75 | 72
Started Protocol Therapy | 3 | 6 | 66 | 66
Eligible | 3 | 6 | 72 | 69
Eligible and Treated | 3 | 6 | 64 | 64
Completed | 3 | 6 | 53 | 49
Not Completed | 0 | 0 | 22 | 23
Not completed — Progressive disease | 0 | 0 | 3 | 3
Not completed — Adverse Event | 0 | 0 | 5 | 4
Not completed — Death | 0 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 3
Not completed — Alternative therapy | 0 | 0 | 0 | 2
Not completed — Other complicating disease | 0 | 0 | 1 | 0
Not completed — Ineligible/never start protocol therapy | 0 | 0 | 11 | 8

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Groups:
- Phase I: The phase I portion of the study was designed to determine the recommended dose for veliparib for the phase II portion of the trial. A total of 9 patients were treated on the phase I study. A total of 3 dose levels of veliparib were planned: 60mg (level 1), 100gm (level 2) and 40mg (level -1). 1 cycle=3 weeks, maximum of 4 cycles.
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II: Arm D (Veliparib) | Phase II: Arm E (Placebo) | Total
Number analyzed (Participants) | 9 | 64 | 64 | 137
Age, Continuous [Median (Full Range); unit: years] | 60 [51 to 78] | 66 [47 to 88] | 64 [45 to 83] | 65 [45 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 30 | 32 | 67
  Male | 4 | 34 | 32 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 5
  White | 8 | 61 | 57 | 126
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose (Phase I)
Description: dose of veliparib which was deemed to be the recommended phase II dose to be administered in the combination with CE for the phase II clinical trial
Time Frame: assessed for a maximum of cycle 1
Population: all eligible and treated patients
Measure: Number; unit: mg
Arm/Group | Phase I
Number analyzed (Participants) | 9
mg | 100

2. Primary Outcome: Progression Free Survival (Phase II)
Description: Profession free survival (PFS) is defined as time from randomization to date of disease progression or death from any cause, whichever occurred first. Patients who had not experienced an event of interest by the time of analysis were censored at the date they were last known to be alive and progression-free. Tumor response was evaluated via Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria, and progression was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, or appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Median PFS was estimated using the Kaplan-Meier method.
Time Frame: Assessed every 3 months for patients < 2 years from registration and every 6 months if patient is 2- 3 years from registration until the date of first documented progression or death. No specific requirements if patient is > 3 years from registration
Population: Eligible and treated patients
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Phase II: Arm D (Veliparib) | Phase II: Arm E (Placebo)
Number analyzed (Participants) | 64 | 64
months
  Overall sample | 6.1 [5.9 to 6.2] | 5.5 [5.1 to 5.7]
  Patients within the male/abnormal LDH stratum: number analyzed (Participants) | 23 | 23
  Patients within the male/abnormal LDH stratum | 6.2 [5.9 to 7.5] | 5.1 [4.3 to 5.5]
  Patients not within the male/abnormal LDH stratum: number analyzed (Participants) | 41 | 41
  Patients not within the male/abnormal LDH stratum | 6.0 [5.8 to 6.3] | 5.6 [5.3 to 6.3]
Statistical Analysis 1: Comparison: Phase II: Arm D (Veliparib) vs Phase II: Arm E (Placebo); The significance test reported here was for treatment arms comparison in patients within the male/abnormal LDH stratum; Test type: Superiority; p < 0.001, Regression, Cox — one-sided p value; adjusted for ECOG performance status, abnormal protein in the Cox proportional hazard model; Hazard Ratio (HR) = 0.34, 80% CI 2-sided [0.22 to 0.51]
Statistical Analysis 2: Comparison: Phase II: Arm D (Veliparib) vs Phase II: Arm E (Placebo); The significance test reported here was for treatment arms comparison in patients not in the male/abnormal LDH stratum; Test type: Superiority; p = 0.18, Regression, Cox — one-sided p value; adjusted for ECOG performance status, abnormal protein in the Cox proportional hazard model; Hazard Ratio (HR) = 0.81, 80% CI 2-sided [0.60 to 1.09]
Statistical Analysis 3: Comparison: Phase II: Arm D (Veliparib) vs Phase II: Arm E (Placebo); If there was a significant treatment-by-stratification factor interaction, the results would be reported separately for each stratum. Significance was defined as the p value was less than 0.05; Test type: Superiority; p = 0.028, Regression, Cox — p value for the interaction by treatment and stratification factor

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as time from randomization to death from any cause. Median OS was estimated using the Kaplan-Meier method.
Time Frame: Assessed every 3 months for patients < 2 years from registration and every 6 months if patient is 2- 3 years from registration until the date of death. No specific requirements if patient is > 3 years from registration
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: Arm D (Veliparib) | Phase II: Arm E (Placebo)
Number analyzed (Participants) | 64 | 64
months | 10.3 [8.9 to 12.0] | 8.9 [8.3 to 11.3]
Statistical Analysis 1: Comparison: Phase II: Arm D (Veliparib) vs Phase II: Arm E (Placebo); Test type: Superiority; p = 0.17, Regression, Cox; stratified on the stratification factors used for randomization; Hazard Ratio (HR) = 0.83, 80% CI 2-sided [0.64 to 1.07]

4. Secondary Outcome: Overall Response Rate (ORR)
Description: Tumor response was evaluated using Response Evaluation Criteria In Solid Tumors (RECIST) v1.1. Complete response (CR) was defined as disappearance of all target lesions. Partial response (PR) was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Overall response rate= (CR+PR)/all eligible and treated patients
Time Frame: assessed every 6 weeks while on study, then every 3 months for patients < 2 years from registration and every 6 months if patient is 2- 3 years from registration.
Population: Eligible and treated patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Phase II: Arm D (Veliparib) | Phase II: Arm E (Placebo)
Number analyzed (Participants) | 64 | 64
percentage of patients | 72 [59 to 82] | 66 [53 to 77]

5. Other Pre Specified Outcome: Neurotoxicity Total Score Change Between Baseline and 3 Months After Treatment Start
Description: Neurotoxicity total score was measured by the 11 items in the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-Ntx) questionnaire. Each item was scored from 0-4. The severity of neurotoxicity was measured by the total score of the 11 items, ranged from 0 to 44. Lower values of the FACT/GOG-Ntx neurotoxicity total score indicate higher neurotoxicity.
Time Frame: assessed at baseline and 3 months after treatment initiation
Population: eligible and treated patients who had neurotoxicity data at both baseline and 3 months assessments
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase II: Arm D (Veliparib) | Phase II: Arm E (Placebo)
Number analyzed (Participants) | 58 | 45
units on a scale | -0.1 (4.8) | -1.8 (6.4)
Statistical Analysis 1: Comparison: Phase II: Arm D (Veliparib) vs Phase II: Arm E (Placebo); Test type: Superiority; p = 0.13, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Assessed every cycle (1 cycle= 21 days) while on treatment and for 30 days after the end of treatment
Groups:
- Phase I: Arm B (Dose Level 2): The phase I portion of the study was designed to determine the recommended dose for veliparib for the phase II portion of the trial. A total of 9 patients were treated on the phase I study. A total of 3 dose levels of veliparib were planned: 60mg (level 1), 100gm (level 2) and 40mg (level -1). 1 cycle=3 weeks, maximum of 4 cycles.
Arm/Group | Phase I: Arm A (Dose Level 1) | Phase I: Arm B (Dose Level 2) | Phase II: Arm D (Veliparib) | Phase II: Arm E (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 51/66 | 54/66
Serious Adverse Events (participants affected / at risk) | 2/3 | 6/6 | 47/66 | 40/66
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 63/66 | 62/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Arm A (Dose Level 1) (N=3) | Phase I: Arm B (Dose Level 2) (N=6) | Phase II: Arm D (Veliparib) (N=66) | Phase II: Arm E (Placebo) (N=66)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 12 | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0
Heart failure (Cardiac disorders) | 0 | 1 | 0 | 0
Death NOS (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 0 | 2
Fever (General disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Duodenal infection (Infections and infestations) | 0 | 0 | 1 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 4 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 6 | 21 | 14
Platelet count decreased (Investigations) | 0 | 2 | 0 | 1
Weight loss (Investigations) | 0 | 0 | 0 | 1
White blood cell decreased (Investigations) | 1 | 5 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 3 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Arm A (Dose Level 1) (N=3) | Phase I: Arm B (Dose Level 2) (N=6) | Phase II: Arm D (Veliparib) (N=66) | Phase II: Arm E (Placebo) (N=66)
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 6 | 12 | 16
Chills (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 5 | 3 | 0
Fever (General disorders) | 0 | 1 | 0 | 0
Infusion related reaction (General disorders) | 1 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 4 | 42 | 35
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 6
Constipation (Gastrointestinal disorders) | 0 | 3 | 3 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 4 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 3 | 2 | 0 | 1
Platelet count decreased (Investigations) | 1 | 5 | 0 | 0
White blood cell decreased (Investigations) | 3 | 3 | 0 | 0
Investigations - Other, specify (Investigations) | 1 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less